CLINICAL TRIAL: NCT04546542
Title: Analysis of Hydroxychloroquine Blood Levels in Patients With Primary Sjögren Syndrome and Possible Correlation With the Disease Activity
Brief Title: Hydroxychloroquine Blood Levels in Primary Sjögren Syndrome Patients
Acronym: 1ASSJHCQ
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1ASSJ
Record Dates: First submitted 2020-08-27; First posted 2020-09-14 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pSS patients under Hydroxychloroquine (HCQ) 2016-AAO dose: Patients under Hydroxychloroquine (HCQ) 2016-American Academy of ophtalmology (AAO) dose will have HCQ blood levels, disease activity and adherence evaltuated at study entry and before 3 and 6-months.
  Interventions: Other: Parallel Assignment

INTERVENTIONS:
Other: Parallel Assignment — We will evaluate 75 patients with pSS (Consenso Americano-europeu de 2002 / EULAR/ACR Classification Criteria, 2016) of both sexes at baseline and 6-months
  Other Names: pSS

SUMMARY:
Introduction. Primary Sjögren's syndrome (pSS) is an autoimmune disease characterized by chronic inflammatory infiltration of the salivary and lacrimal glands causing dry eye and mouth. Multiple systemic manifestations can also occur. Hydroxychloroquine (HCQ), an antimalarial immunomodulator, has been used for the treatment of arthralgias, myalgia and constitutional symptoms resulting from pSS. However, there are no studies that evaluated whether blood levels of HCQ could influence in the therapeutic response, as has been reported in systemic lupus erythematosus (SLE).

Objectives. Analyze in patients with pSS receiving HCQ as part of their treatment: blood levels of HCQ; adherence using a questionnaire versus blood levels and the possible correlation of blood levels with the disease activity score in a cross-sectional evaluation followed by a longitudinal six-month assessment.

Patients and methods. Observational cross-sectional evaluation followed by a six-month longitudinal assessment, including patients with pSS receiving HCQ for at least 3 months at study admission. Patients will be evaluated clinically and the HCQ blood level measured at the beginning of the study (T0), at 3 months (T3), and at 6 months (T6). As there are no previous studies on blood levels of HCQ in patients with pSS, the sample of 75 patients was calculated based on the percentage of these patients currently using HCQ in our service (nearly 50%) and in the number of patients in current follow-up (about 150). We will evaluate 75 adult patients with pSS according to the classification criteria of the American-European Consensus Group 2002 and/or the American College of rheumatology (ACR) and the European League Against Rheumatism (EULAR) 2016, of both sexes and followed up regularly at the Sjögren Syndrome outpatient Clinic of the Rheumatology Service of "Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (HCFMUSP)". The following will be used in the clinical evaluation: the xerostomia Inventory; the xerophthalmia questionnaire - Ocular Surface Disease Index (OSDI); the EULAR Sjögren Syndrome Reported Index (ESSPRI); the EULAR Sjögren Syndrome Disease Activity Index (ESSDAI); the Sjögren's Syndrome Disease Damage Index (SSDDI); the non-stimulated and stimulated salivary flow. Blood levels of HCQ will be measured by high performance liquid chromatography and tandem mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* pSS according to the classification criterias
* Who have been receiving HCQ for at least 3 months before study entry
* Patients who agree to participate in the study, according to the signing of the Free and Informed Consent Term (ICF).

Exclusion Criteria:

* Present other associated systemic autoimmune diseases, such as rheumatoid arthritis, systemic lupus erythematosus, systemic sclerosis, demato/polymyositis, mixed connective tissue disease, spondyloarthritis, primary biliary cholangitis and autoimmune hepatitis;
* Present a previous history of radiotherapy of the head and neck, positive serologies for HIV, hepatitis B and C, sarcoidosis, graft versus host disease and IgG4-related disease;
* Use of drugs that can interact with HCQ or interfere in HCQ blood levels (tamoxifen, antacids and digoxin), alcoholism, current infections, liver and heart failure, dialysis, severe chronic renal failure (serum creatinine ≥3 mg/dL) and pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pSS patients according to the classification criterias regularly followed at outpatient clinic, Rheumathology division of Hospital das Clinicas da Universidade de Sao Paulo
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline of HCQ blood levels at 3 and 6 months | Baseline, 3 and 6 months
  Hydroxychloroquine blood levels will be measure using liquid chromatography tandem Mass Spectrometry (LC-MS/MS), as previously described (PEDROSA et al., 2020).

SECONDARY OUTCOMES:
HCQ adherence in pSS patients | Baseline, 3 and 6 months
  Will be analysed the possible correlation between MTA (measure for treatment adhernce - a quesionnaire of adherence) score and HCQ blood levels em ng/mL (using liquid chromatography tandem Mass Spectrometry (LC-MS/MS), as previously described (PEDROSA et al., 2020). For SLE patients, adherence by HCQ blood levels is defined when HCQ blood levels are >500 ng/mL, this value in pSS patients will be estimated using this 2 assessements
Disease activity in pSS patients | Baseline, 3 and 6 months
  We will evaluate the disease activity in pSS patients and correlate if HCQ blood levels can predict risk of disease acrivity

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Rheumatology Division of Hospital das Clínicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pedrosa TN, Pasoto SG, Aikawa NE, Yuki EF, Borba EF, Filho JCF, Carricondo PC, Zanetti CB, Conde PG, Duarte NJ, Fontoura N, Romano P, Carvalho VM, Silva CA, Bonfa E. Understanding the dynamics of hydroxychloroquine blood levels in lupus nephritis. Lupus. 2020 May;29(6):560-568. doi: 10.1177/0961203320912832. Epub 2020 Mar 19. No abstract available. PMID 32192398
- [Result] Cankaya H, Alpoz E, Karabulut G, Guneri P, Boyacioglu H, Kabasakal Y. Effects of hydroxychloroquine on salivary flow rates and oral complaints of Sjogren patients: a prospective sample study. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Jul;110(1):62-7. doi: 10.1016/j.tripleo.2010.02.032. PMID 20610299
- [Result] Yavuz S, Asfuroglu E, Bicakcigil M, Toker E. Hydroxychloroquine improves dry eye symptoms of patients with primary Sjogren's syndrome. Rheumatol Int. 2011 Aug;31(8):1045-9. doi: 10.1007/s00296-010-1415-4. Epub 2010 Mar 23. PMID 20309693